CLINICAL TRIAL: NCT01607463
Title: The Effect of Transcutaneous Electrical Nerve Stimulation on Pain During Venous Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Younghoon Jeon, Anesthesiology and Pain Medicine, Kyungpook National University Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: KNUH 2012-04-014-001
Record Dates: First submitted 2012-05-22; First posted 2012-05-30 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Cannulation Pain
Keywords: pain; transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- active TENS group (Experimental): Two electrodes were attached to the radial side of dominant forearm. In the active TENS group, TENS was delivered via two electrodes on the venous cannulation site
  Interventions: Procedure: Transcutaneous electrical nerve stimulation (Empi, USA)
- Placebo group (Placebo Comparator): Two electrodes were attached to the radial side of dominant forearm. In the placebo group the TENS device had no current output although the power "on" indicator light remained active.
  Interventions: Procedure: Transcutaneous electrical nerve stimulation (Empi, USA)

INTERVENTIONS:
Procedure: Transcutaneous electrical nerve stimulation (Empi, USA) — In the active TENS group, TENS at 80 pulsed currents per second (PPS) with a pulse duration of 200 μs were delivered for 20 minutes. Current amplitude was slowly increased until a level was reached that participants reported was the maximum level they could tolerate below pain threshold without noticeable muscle contraction and maintained this intensity.
  Arms: active TENS group
Procedure: Transcutaneous electrical nerve stimulation (Empi, USA) — In the placebo group the TENS device had no current output although the power "on" indicator light remained active.
  Arms: Placebo group

SUMMARY:
The purpose of this study was to investigate whether transcutaneous electrical nerve stimulation (TENS) could reduce pain during cannulation of vein.

DETAILED DESCRIPTION:
One hundred patients were allocated randomly to two groups: In the active TENS group TENS was delivered via two electrodes on the venous cannulation site (radial side of the wrist of dominant forearm) 20 min prior to venous cannulation and control group received placebo (no current) TENS. Venous cannulation with a 22 gage cannula was performed. During venous cannulation the pain intensity (0 = no pain, 10 = worst pain imaginable) was measured. Any side effects during study periods were recorded

ELIGIBILITY:
Inclusion Criteria:

* outpatients who underwent plastic surgery

Exclusion Criteria:

* concomitant sedative or analgesic medication,
* neurological disease.
* all patients with potentially dangerous internal diseases (American Society of Anesthesiologists' physical status > 3).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The effect of transcutaneous electrical nerve stimulation on pain during venous cannulation | one minute after cannulation
  One hundred patients were allocated randomly to two groups: In the active TENS group TENS was delivered via two electrodes on the venous cannulation site (radial side of the wrist of dominant forearm) 20 min prior to venous cannulation and control group received placebo (no current) TENS. Venous cannulation with a 22 gage cannula was performed. One minute after venous cannulation the pain intensity (0 = no pain, 10 = worst pain imaginable) was measured. Any side effects during study periods were recorded

CONTACTS AND LOCATIONS:
Overall Officials: Younghoon Jeon, Dr, Principal Investigator — 2. Anesthesiology and Pain Medicine, Kyungpook National University Hospital

REFERENCES:
- [Derived] Kim S, Park K, Son B, Jeon Y. The effect of transcutaneous electrical nerve stimulation on pain during venous cannulation. Curr Ther Res Clin Exp. 2012 Sep;73(4-5):134-9. doi: 10.1016/j.curtheres.2012.05.001. PMID 24653515